CLINICAL TRIAL: NCT04112680
Title: The Contagious Misinformation Trial: Debunking Prevalent Misinformation About an Infectious Disease Through Audio Dramas in Freetown, Sierra Leone
Brief Title: Contagious Misinformation Trial
Acronym: CMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Nordenstedt, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CMT2019
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Misinformation
Keywords: Misinformation; Communication; Infectious diseases
MeSH Terms: conditions — Communication; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Interventional study, with 3 arms (2 intervention groups, 1 control group) to test communication elements of audio dramas aiming to counter prevalent belief in misinformation about an infectious disease in Freetown, Sierra Leone
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant will not know the group they are assigned to, as all groups (also the control group) will receive audio messages.
  The investigator and outcomes assessors will only be handed an anonymised data set.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): Audio messages in this group are focussed on providing a Plausible Alternative to the misinformation
  Interventions: Behavioral: Debunking Misinformation through Audio Dramas
- Intervention group 2 (Experimental): Audio messages in this group focus on Avoiding the Misinformation and instead only provide the correct information
  Interventions: Behavioral: Debunking Misinformation through Audio Dramas
- Control group (Placebo Comparator): Audio messages in this control group are on a different topic
  Interventions: Behavioral: Control group audio jingles

INTERVENTIONS:
Behavioral: Debunking Misinformation through Audio Dramas — The audio dramas (one drama of 4 episodes per intervention group), aim to debunk misinformation about an infectious disease. The content of the two dramas differ in the two groups; in intervention group 1, the drama will state the misinformation and provide a plausible alternative, delivered through a trusted source, in line with world views. In intervention group 2, the audio drama will avoid mentioning the misinformation and instead only state the correct information about the infectious disease
  Arms: Intervention group 1; Intervention group 2
Behavioral: Control group audio jingles — The control group will receive audio jingles about exclusive breastfeeding
  Arms: Control group

SUMMARY:
In the Contagious Misinformation Trial the investigators aim to debunk prevalent misinformation about an infectious disease using two evidence-based methods of debunking. The two debunking methods are packaged in two audio dramas of 4 episodes each, which will be sent to the WhatsApp of participants who are randomised to intervention group 1 or 2. The control group will receive audio messages about a different topic. The primary outcome is the reduction in belief in two misinformation statements about the infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Living in Freetown
* In possession of a mobile phone that has WhatsApp
* Fluent in Krio

Exclusion Criteria:

* Deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Change in the belief in misinformation | Up to 2 months
  The change in the belief in misinformation will be measured through Yes/No questions in the baseline and follow-up surveys. Using logistic regression models, the prevalence of the belief in misinformation about 2 aspects of an infectious disease compared to the control group will be analysed using an intention-to-treat and per-protocol analysis

SECONDARY OUTCOMES:
Inadvertent promotion of misinformation: the backfire effect | Up to 2 months
  To test whether the interventions might inadvertently have promoted the belief in misinformation, the same yes/no questions as the primary outcome will be used in ordinal logistic regression models to analyse if the there has been a backfire effect in the intervention groups, compared to the control group.
As treated analysis of primary outcomes | Up to 2 months
  The Yes/No questions of the primary outcomes will be tested in an as-treated analysis. The investigators will only include participants who can correctly recall the basic storylines of the audio messages.
Knowledge about preventive methods | Up to 2 months
  Using an open question, asking the respondent to name up to 3 preventive methods, a score will be created. For every correct answer, the participants gets a point, and one point is subtracted for every wrong answer; leading to a potential score of -3 to +3. Ordinal logistic regression models will be fitted to compare the scores of the intervention groups with the control group.
Health-related discussions among family/friend | Up to 2 months
  The question asking whether the participant has discussed the content of the audio messages will be used for this analysis, together with the question about how often the participant discussed health issues with family/friends. Logistic regression models will be fitted to test whether the interventions have influenced health-related discussions with family or friends, as compared to the control group.
Method of administration | Up to 2 months
  To understand if the intervention works outside of WhatsApp, 60 additional people will be recruited who do not have WhatsApp. Participants will instead be called and listen to the audio dramas on the phone; 30 will listen to the audio drama of intervention group 1 and 30 will listen to the audio drama of intervention group 2. The two primary outcomes will be analysed similar to the primary outcome analysis (ITT and per protocol) among the 2 groups and compared to the control group, as well as to their equivalent group of respondents with WhatsApp.
Differences in self-efficacy | Up to 2 months
  Participants will answer 3 questions about their perceived self-efficacy on 3 specific preventive behaviours. Answers are on a 5-item scale: from not at all true to exactly true. Ordinal logistic regression models will be specified to test whether the interventions had an influence on people's self-efficacy about three specific preventive behaviours, compared to the control group.
Risk perception & preventive methods | Up to 2 months
  Risk perception about the infectious disease will be measured with a question that asks how likely it is that the participants gets the disease in the next year. A question which asks what kind of actions the participants has undertaken, or is planning to undertake, to prevent infection with the disease - will be used to assess if and what kind of actions are taken. Several analyses will be carried out to test whether the intervention influenced risk perception and preventive methods. Furthermore, analyses will be carried out to determine if the a change in risk perception influenced preventive methods.
Objective versus subjective learning | Up to 2 months
  In the follow-up survey, there is a question asking if the participant feels like he/she learned from the audio messages (yes/no question). A Chi-Square analysis will be done to determine whether those who feel like they learned also learned objectively, using the two primary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Nordenstedt, MD PHD, Principal Investigator — Karolinska Institutet
Locations (1):
- Focus1000, Freetown, Western Area, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
After publication of the primary analysis and study results, the anonymised data will be published in a public repository
Supporting Information: SAP, ICF
Time Frame: January 2022

REFERENCES:
- [Derived] Winters M, Oppenheim B, Sengeh P, Jalloh MB, Webber N, Pratt SA, Leigh B, Molsted-Alvesson H, Zeebari Z, Sundberg CJ, Jalloh MF, Nordenstedt H. Debunking highly prevalent health misinformation using audio dramas delivered by WhatsApp: evidence from a randomised controlled trial in Sierra Leone. BMJ Glob Health. 2021 Nov;6(11):e006954. doi: 10.1136/bmjgh-2021-006954. PMID 34758970

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04112680/SAP_000.pdf
  • Study Protocol (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04112680/Prot_001.pdf